CLINICAL TRIAL: NCT05400733
Title: Prandial Metabolic Phenotype in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Professor, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 83 - Pulse Feeding
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Protein Metabolism
Keywords: prandial
MeSH Terms: interventions — Amino Acids, Essential; Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy male older adults (Other): Healthy male older adults
  Interventions: Dietary Supplement: Total Amino Acids; Dietary Supplement: Essential Amino Acids; Dietary Supplement: Essential Amino Acids + Hydroxy-methylbutyric acid (HMB); Dietary Supplement: Essential Amino Acids + Leucine; Dietary Supplement: Essential Amino Acids High; Dietary Supplement: Placebo Water
- Healthy female older adults (Other): Healthy female older adults
  Interventions: Dietary Supplement: Total Amino Acids; Dietary Supplement: Essential Amino Acids; Dietary Supplement: Essential Amino Acids + Hydroxy-methylbutyric acid (HMB); Dietary Supplement: Essential Amino Acids + Leucine; Dietary Supplement: Essential Amino Acids High; Dietary Supplement: Placebo Water

INTERVENTIONS:
Dietary Supplement: Total Amino Acids — Histidine, Isoleucine, Leucine, Lysine, Methionine, Phenylalanine, Threonine, Tryptophan, Valine, Alanine, Arginine, Aspartate, Cystine, Glutamine, Glutamate, Glycine, Proline, Serine, Tyrosine. All supplements are commercially available.
Dietary Supplement: Essential Amino Acids — Histidine, Isoleucine, Leucine, Lysine, Methionine, Phenylalanine, Threonine, Tryptophan, Valine. All supplements are commercially available.
Dietary Supplement: Essential Amino Acids + Hydroxy-methylbutyric acid (HMB) — Histidine, Isoleucine, Leucine, Lysine, Methionine, Phenylalanine, Threonine, Tryptophan, Valine, HMB. All supplements are commercially available.
Dietary Supplement: Essential Amino Acids + Leucine — Histidine, Isoleucine, Leucine, Lysine, Methionine, Phenylalanine, Threonine, Tryptophan, Valine, Extra leucine. All supplements are commercially available.
Dietary Supplement: Essential Amino Acids High — Histidine, Isoleucine, Leucine, Lysine, Methionine, Phenylalanine, Threonine, Tryptophan, Valine. All supplements are commercially available.
Dietary Supplement: Placebo Water — Water

SUMMARY:
Previous studies suggest that changes in metabolism due to the effects of aging might serve as a potential for therapeutic agents. The investigating lab developed a pulse method combining multiple stable isotopes to study multiple metabolic pathways in the same individual simultaneously. By measuring whole-body metabolism in a large group of older adults, the investigators may be able to unravel age-related deterioration in protein turnover (synthesis and breakdown) that contributes to impaired functional capacity. Metabolic profiles could explain differences in pathways in the aging process with special interest in metabolism of amino acids as they have been associated with aging-related disorders.

DETAILED DESCRIPTION:
The study involves 1 screening visits of approximately 3 hours and 6 study days of approximately 8 hours.

Subjects will be asked to arrive in the fasted state on all study days. Fasting prior to screening is not required. On the screening day, body weight, height, and body composition by Dual-energy X-ray absorptiometry (DXA) will be measured. In addition, The Six-Minute Walk Test (6MWT) and skeletal muscle function tests will be assessed at the end of each screening visit.

Each study visit will begin with vital signs. Before administration of the feeding or the tracer solution, baseline blood will be collected for measurement of the natural enrichment of metabolites. After the baseline sample is collected, feeding will begin and will be followed by tracers of several compounds that may be administered by IV pulse.

Next, the subjects will be fed one of six liquid nutritional supplement every 20 minutes for 6 hours. The liquid nutrition supplement will target the amino acid formulation in the following meals (1) total amino acid, (2) Essential Amino Acids (EAA), (3) EAA + -hydroxy -methylbutyric acid (HMB), (4) EAA + leucine (LEU), (5) EAA high, and (6) Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60-80, inclusive
* Stable body-weight (± 5%) for the past 3 months
* Subject is judged to be in satisfactory health based on medical history, physical examination, and laboratory screening evaluations.
* Ability to walk, sit down and stand up independently or with walking mobility aids
* Ability to lie in supine or elevated position for up to 7 hours
* Willingness and ability to comply with the protocol

Exclusion Criteria:

* Established diagnosis of current malignancy
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Use of short course of oral corticosteroids within 4 weeks preceding study day
* (Possible) pregnancy
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* Already enrolled in another clinical trial and that clinical trial interferes with participating in this study
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Feeding related changes in whole-body protein and amino acid metabolism | up to 6 hours
  Whole-body production rate measured after stable tracer administration

CONTACTS AND LOCATIONS:
Locations (1):
- Human Clinical Research Facility, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared upon request for up to 6 years beyond completion of the trial based on methods/proposal approved by both parties' institutional review committees. Individual participant data that underlie the results of the trial may be shared after de-identification (text, tables, figures, and appendices). Additional documents available per request include: study protocol, statistical analysis plan, and informed consent. Requests should be directed to Dr. Marielle Engelen (mpkj.engelen@ctral.org).

REFERENCES:
- [Derived] Deutz NEP, Knezek SB, Engelen MPKJ. A novel pulse tracer method to estimate the relationship between amino acid meal composition and its intracellular disposal. Clin Nutr. 2025 Dec;55:196-207. doi: 10.1016/j.clnu.2025.10.002. Epub 2025 Oct 22. PMID 41260190